CLINICAL TRIAL: NCT02107885
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled Single Ascending Dose Study to Assess Safety, Tolerability and Pharmacokinetics of DS-1971a in Healthy Male Subjects
Brief Title: Single Ascending Dose Study Using DS-1971 to Assess Safety, Tolerability, and Pharmacokinetics in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DS1971-A-E101
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2014-10

CONDITIONS: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS-1971 (Experimental): single ascending dose of 5mg, 10mg, 30mg, 90mg, 250mg, 500mg, 1000mg, 1500mg.
  Interventions: Drug: DS-1971
- placebo (Placebo Comparator): placebo matching each of the DS-1971 dosages.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-1971 — 6 subjects in each group will receive DS-1971.
  Arms: DS-1971
Drug: placebo — 2 subjects in each group will receive placebo.
  Arms: placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled and ascending single dose study. It is hypothesised that single oral doses of DS-1971a within the planned dose range will be safe and well tolerated by healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18-45 years.
* A body mass index (BMI or Quetlet index) in the range 18-30 kg/m^2, inclusive, and weighing between 50 and 100 kg at screening.

Body Mass Index (BMI) =weight[kg] / (height [m])^2

* Willing to use a reliable method of contraception and not donate sperm during the study, and for 4 months afterwards.
* Sufficient intelligence to understand the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with requirements of, the entire study.
* Willing to give written consent to participate in the study after reading the ICF, and after having the opportunity to discuss the study with the Investigator or his delegate.
* Willing to give written consent to have his data entered into The Over-volunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings, or laboratory values that could interfere with the objectives of the study or compromise the safety of the subject.
* Presence or history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* History of serious reaction to any medicine.
* Presence or history of malignant disease.
* Acute or chronic infectious disease, including HIV, HBV or HCV infection.
* Surgery (e.g. stomach bypass) or medical condition that might affect how the body handles or absorbs medicines.
* Significant illness within 4 weeks before the dose of trial medication.
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of trial medication.
* Abnormal ECG waveform morphology at screening that would preclude accurate measurement of the QT interval duration.
* QTcF interval duration > 430 msec, obtained as an average from the 3 ECG measurements on the triplicate screening ECGs.
* Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m^2MDRD] equation).
* Use of any prescription or OTC medications known to be strong inhibitors or strong inducers of CYP enzymes (also known as CYP P450 enzymes) during the 30 days before the dose of trial medication; use of any other prescription or OTC medicine including vitamins or herbal remedies like St John's wort, with the exception of acetaminophen (paracetamol), during the 7 days before the dose of trial medication.
* Consumption of grapefruit, grapefruit juice or Seville oranges within 10 days before the dose of trial medication, or unwilling to abstain from consuming them throughout the study.
* Consumption of food or beverages containing caffeine or xanthine within 24 h before admission on Day -1, or unwilling to abstain from consuming them for 3 days after receiving the trial medication.
* Loss of more than 400 mL blood during the 3 months before the study.
* Donation of blood, plasma, platelets, or any other blood components during the 3 months before the study, or unwilling to abstain from doing so during the study and for 3 months after receipt of trial medication.
* Abuse of drugs or alcohol during the 2 years before the dose of trial medication, or intake of more than 21 units of alcohol weekly.
* Use of tobacco products or nicotine-containing products during the 3 months before the dose of trial medication.
* Evidence of drug or alcohol abuse at screening or admission.
* Likely possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by GP to the volunteer entering the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
safety and tolerability adverse events | 20 days after dose
  determine number, type, and severity of adverse events
safety and tolerability physical exam | 20 days after dose
  determine adverse changes in vital signs, ECG.
safety and tolerability laboratory blood and urine tests | from day 1 through 20 days after dose
  determine adverse changes in laboratory safety tests of blood (biochemistry and haematology) and urine.

SECONDARY OUTCOMES:
plasma concentration AUC | day 4
  concentration in blood measured as Area under the curve (AUC)
maximum blood concentration | day 4
  Cmax
time of maximum blood concentration | day 4
  T_max
half-life of drug in body | day 4
  T_1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/